CLINICAL TRIAL: NCT01808677
Title: Registry Study of Thoracic Reirradiation for Non-Small Cell Lung Cancer (NSCLC) Utilizing Proton Beam Therapy or Intensity Modulated Radiation Therapy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA11-1193
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Thoracic reirradiation; Proton beam therapy; PBT; Intensity modulated radiation therapy; IMRT; Registry; Data
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracic Reirradiation Registry: Data collection on patients being treated with thoracic reirradiation with PBT or IMRT for NSCLC, with or without chemotherapy.
  Interventions: Other: Thoracic Reirradiation Registry

INTERVENTIONS:
Other: Thoracic Reirradiation Registry — Data collected in the registry includes patient characteristics/demographics, disease characteristics, treatment details (radiation, chemotherapy, surgery, etc.), toxicity rates, and survival outcomes.

SUMMARY:
The goal of this research study is to learn more about the safety of treating NSCLC with reirradiation using standard methods and to look for ways to lessen side effects and improve therapy. Reirradiation is when radiation is given to an area of the body that has previously received a full dose of radiation.

DETAILED DESCRIPTION:
If you agree to take part in this study, data will be recorded during your therapy. The data to be recorded will include your medical history, the disease, treatments you have received and how you have responded to any treatments, as well as any side effects you may have had.

The data will be stored on a password-protected computer at MD Anderson for use in future research related to cancer.

Your data will be given a code number. No identifying information will be directly linked to your data. Only the researcher in charge of this study will have access to the code numbers and be able to link the data to you. This is to allow medical information related to your data to be updated as needed. Other researchers using your data will not be able to link this data to you.

Length of Study:

After you sign this consent form, your active participation on this study will be over.

This is an investigational study.

Up to 120 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. History of previous histologically or cytologically documented NSCLC, stage I-IV.
2. Prior course of radiation therapy or concurrent chemoradiation at least 1 month prior to the current course of radiation therapy.
3. Patients eligible to receive a second course of radiation therapy to the thorax, at the discretion of the treating physician.
4. Patients receiving concurrent chemotherapy or targeted agents will be eligible for this protocol.

3.2 Exclusion Criteria:

1. Life expectancy<3 months
2. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated with thoracic reirradiation with PBT or IMRT for NSCLC, with or without chemotherapy at UT MD Anderson Cancer Center in Houston, Texas.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of High-Grade Toxicity | 5 years
  Primary objective to assess the prevalence of high-grade toxicity in patients being treated with thoracic reirradiation with proton beam therapy (PBT) or intensity modulated radiation therapy (IMRT) for non-small cell lung cancer (NSCLC), with or without chemotherapy. High-grade toxicity defined as CTCAE v4.0 Grade 3 or higher toxicity, or CTCAE v4.0 grade 4 or higher toxicity of the esophagus. Data collected from 1/2/2012 to 1/31/2017. High-grade toxicity rate and its corresponding 95% confidence interval provided at end of study. Logistic regression model used to assess the association between prognostic factors such as total dose to normal tissue structures, time since initial course of RT, failure in same lobe of the lung, failure in nodal regions, and central vs. peripheral location and high-grade toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gomez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org